CLINICAL TRIAL: NCT05551130
Title: Is There a Possibility That Bulk Fill Glass Hybrid Restorative Materials Could Replace Composite Resins in Treating Permanent Teeth? : A Randomized Controlled Clinical Trial
Brief Title: Could Bulk Fill Glass Hybrid Restorative Materials Replace Composite Resins in Treating Permanent Teeth?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hazal Özer, Assist. Prof., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/332
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Dental Restoration Failure of Marginal Integrity
Keywords: Composite Resins; Clinical Trial; Glass Ionomer Cements; Permanent Dental Restoration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equia Group (Active Comparator): Equia system bulk fill glass hybrid material
  Interventions: Other: Restoration
- Charisma Group (Active Comparator): Charisma Smart universal composite resin
  Interventions: Other: Restoration

INTERVENTIONS:
Other: Restoration — Restorations completed with these materials.
  Other Names: Restorative Interventions

SUMMARY:
The aim of this study is to compare the clinical and radiographic efficacy of Equia system bulk fill glass hybrid material with composite resins in the permanent restoration of pediatric patients' permanent teeth.

DETAILED DESCRIPTION:
The study included 44 pediatric patients aged 8 to 16 years who applied to the Pedodontics Department of the Necmettin Erbakan University Faculty of Dentistry. The groups were formed as symmetrical teeth in the same patient using the split-mouth design. The study included class I caries lesions of 144 permanent teeth, 72 of which were restored with the Equia system bulk fill glass hybrid material [Equia Forte HT+Equia Forte Coat (GC, Co, Tokyo, Japan)] and 72 with the Charisma Smart universal composite resin (Kulzer, Gmbh, Hanau, Germany) + Clearfil SE Bond (Kuraray, Noritake, Sakazu, Okayama). Evaluations were performed clinically and radiographically by 2 physicians in the 2nd week, 3rd month, 6th month, and 12th month and the results were recorded. Clinical evaluation was carried out using modified USPHS criteria. Obtained data were statistically analyzed using Kendall's W test and Cochran's Q test for the comparison within the group, and the Chi-Square test for the comparison between the groups.

ELIGIBILITY:
Inclusion Criteria:

* The patient has no systemic disease
* The patient should have good periodontal status
* Teeth to be restored should be symptomless and vital
* Teeth to be restored should have proximal contacts on both mesial and distal surfaces and be in occlusion with the antagonist teeth
* Teeth that have class II caries lesions in external and middle 1/3 of dentine thickness radiographically

Exclusion Criteria:

* Xerostomia and bruxism;
* Absence of adjacent and antagonist teeth;
* Extremely poor oral hygiene, severe or chronic periodontitis;
* Teeth that have any restoration, endodontic treatment, periodontal and periapical pathology.
* The patients who are undergoing orthodontic treatment

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
marginal adaptation | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
marginal discoloration | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
color match | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
surface texture | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
secondary caries | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
postoperative sensitivity | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie
retention | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie

SECONDARY OUTCOMES:
anatomic form | 2 weeks-12 months
  According to the amended USPHS (United States Public Health Service) criteria, a direct clinical evaluation was conducted.
  The scale:
  Alfa Bravo Charlie

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Abakli Inci, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The research will be published soon.